CLINICAL TRIAL: NCT00058045
Title: A Phase I Study Of Low-Dose Subcutaneous Interleukin 2 (IL-2) And Stem Cell Factor (r-metHuSCF) For Patients With AIDS And AIDS-Associated Malignancy
Brief Title: Interleukin-2 and Stem Cell Factor in Treating Patients With AIDS or AIDS-Related Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: RP 99-11; RPCI-RP-9911
Record Dates: First submitted 2003-04-07; First posted 2003-04-09 (Estimated); Last update posted 2013-01-31 (Estimated); Status verified 2013-01

CONDITIONS: Lymphoma
Keywords: AIDS-related peripheral/systemic lymphoma
MeSH Terms: conditions — Lymphoma | interventions — aldesleukin; Stem Cell Factor

INTERVENTIONS:
Biological: aldesleukin
Biological: recombinant human stem cell factor

SUMMARY:
RATIONALE: Interleukin-2 may stimulate a person's white blood cells to kill cancer cells. Stem cell factor may increase the number of immune cells found in bone marrow or peripheral blood and may help a person's immune system recover from the side effects of cancer therapy.

PURPOSE: Phase I trial to study the effectiveness of combining interleukin-2 with stem cell factor in treating patients who have AIDS or AIDS-related cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the safety and toxicity of low-dose interleukin-2 and stem cell factor in patients with AIDS or AIDS-related malignancies.
* Determine the immune status of patients treated with this regimen.

OUTLINE: This is a multicenter, dose-escalation study of stem cell factor.

Patients receive interleukin-2 (IL-2) subcutaneously (SC) six days a week and stem cell factor SC three times a week for 8 weeks in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of stem cell factor until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. Once the MTD is determined, an additional cohort of 3 patients receives treatment at the MTD.

Patients are followed every 2 weeks for 1 month.

PROJECTED ACCRUAL: A total of 3-18 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of HIV-1 by ELISA, Western blot, polymerase chain reaction, or other documentation
* Must have had 1 of the following AIDS-defining illnesses:

  * Opportunistic infection
  * Opportunistic malignancy (excluding CNS involvement)
  * CD4 T-cell count less than 200/mm^3 (but currently greater than 20/mm^3)
* Receiving antiretroviral therapy
* No concurrent Kaposi's sarcoma

  * Prior Kaposi's sarcoma in complete response allowed

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* Karnofsky 80-100%

Life expectancy

* Not specified

Hematopoietic

* Absolute granulocyte count greater than 1,000/mm^3*
* Hemoglobin at least 10 g/dL*
* Platelet count greater than 50,000/mm^3* NOTE: *Transfusions and growth factors allowed in order to increase or maintain counts

Hepatic

* No major hepatic dysfunction evidenced by encephalopathy, ascites, or varices
* Bilirubin no greater than 2 mg/dL
* INR no greater than 1.5

Renal

* Not specified

Cardiovascular

* No prior angioedema
* No uncontrolled hypertension (i.e., diastolic blood pressure greater than 115 mmHg)
* No unstable angina
* No New York Heart Association class III or IV heart disease
* No congestive heart failure
* No coronary angioplasty within the past 6 months
* No myocardial infarction within the past 6 months
* No uncontrolled atrial or ventricular cardiac arrhythmia

Pulmonary

* No history of seasonal or recurrent asthma within the past 10 years
* No concurrent asthmatic symptoms (e.g., wheezing) related to a current respiratory tract infection

Immunologic

* No prior positive allergy test (skin or radioallergosorbent test) for insect venoms
* No known allergy to E. coli-derived products
* No prior anaphylactic events manifested by disseminated urticaria, laryngeal edema, and/or bronchospasm
* Drug allergies manifested solely by rash and/or urticaria allowed
* No recurrent urticaria (isolated episode of urticaria allowed)
* No other active uncontrolled infection (including one with current symptoms of bronchoconstriction)
* No fever of 38.2° C or higher

  * Fevers due to B symptoms allowed

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No prior or concurrent CNS malignancy
* No poorly controlled diabetes
* No other significant nonmalignant disease
* No other malignancy except those in stable partial response or stable complete response (no evidence of progressive disease for at least 8 weeks after therapy for the malignancy)

PRIOR CONCURRENT THERAPY:

Biologic therapy

* See Hematopoietic in Patient Characteristics
* No prior stem cell factor
* No concurrent interleukin-11 for thrombocytopenia

Chemotherapy

* No concurrent chemotherapy for malignancy

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* Not specified

Other

* No concurrent enrollment on any other protocol utilizing an investigational drug
* No concurrent beta adrenergic blocking agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2002-08; Primary Completion 2003-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zale P. Bernstein, MD, Study Chair — Roswell Park Cancer Institute
Locations (2):
- United States (2):
  - Roswell Park Cancer Institute, Buffalo, New York
  - Arthur G. James Cancer Hospital - Ohio State University, Columbus, Ohio